CLINICAL TRIAL: NCT00005441
Title: Lifestyle Management for Women With CHD and NIDDM
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4370; R29HL050181 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Diabetes Mellitus, Non-insulin Dependent; Postmenopause; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To develop and evaluate a comprehensive lifestyle self-management (CLSM) program (low-fat vegetarian diet, smoking cessation and stress management training) for postmenopausal women with coronary heart disease and Type II (non-insulin dependent) diabetes.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease is the leading cause of death among postmenopausal women. Yet few studies have examined the potential for altering risk factors for coronary heart diseases among postmenopausal women, especially as a result of comprehensive lifestyle changes. A pressing need existed for controlled studies to evaluate the effects of comprehensive lifestyle changes on risks for coronary heart disease among postmenopausal women.

DESIGN NARRATIVE:

The comprehensive lifestyle management program appeared to produce substantial cardiovascular benefits among men but little was known about the behavioral processes through which change occurred. Its generalizability and applicability -- especially for high-risk women --was uncertain. The program was compared to a usual care condition in an initial randomized trial. Outcome measures included patient self-care behaviors and health outcomes (serum lipid profiles, blood pressure, relative weight, and glycemic control). Process measures included self-efficacy, personal health models, perceived stress, social support and problem-solving skills. Subjects participated in the intervention for three years, with gradual fading of the program in the third year to evaluate the long-term effects of the program. Analyses included assessments of between groups differences on physiological risk factors, behavioral (lifestyle) measures and process measures as well as maintenance over time. Based upon the results of this study, the long-term goal was to design a second outcome study in which the revised intervention would be evaluated with a larger sample to determine the relative contribution of adding moderate exercise and the effects on reversal of coronary heart disease.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-04; Primary Completion 1997-10 (Actual); Study Completion 1998-03 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toobert DJ, Glasgow RE, Nettekoven LA, Brown JE. Behavioral and psychosocial effects of intensive lifestyle management for women with coronary heart disease. Patient Educ Couns. 1998 Nov;35(3):177-88. doi: 10.1016/s0738-3991(98)00074-3. PMID 9887850